CLINICAL TRIAL: NCT01181375
Title: Predictive Assays in Cervix Cancer: Assessment of Hypoxia, Interstitial Fluid Pressure, and Tissue and Plasma Biomarkers of Hypoxia (CXTF10)
Brief Title: Predictive Assays In Cervix Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UHN REB 06-0379-CE
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; assay; hypoxia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Hypoxia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Assays on cervical cancer tissue (Experimental)
  Interventions: Other: Tumour Biopsies and Blood Sampling

INTERVENTIONS:
Other: Tumour Biopsies and Blood Sampling — Patients who consent to the tissue part of this study will have Biopsies taken for study purposes at the same time as their routine tumour biopsies . In addition,those who consent to the blood sampling part of the study will have their samples taken assess serum biomarkers of tumour oxygenation.

SUMMARY:
The experiments outlined in this proposal will compare a number of currently available techniques for assessing hypoxia and interstitial fluid pressures in patients with cervix cancer. The aim of these experiments is to establish the relationship of the clinically relevant outcome measures of tumour control and survival following radiation therapy with these biological characteristics of carcinoma of the cervix relevant to tumour hypoxia. These characteristics will be assessed in patients undergoing treatment using techniques which have reached an appropriate level of development for clinical evaluation and aim to determine the best technique for determining these parameters of the tumour microenvironment. A number of novel strategies directed at the microenvironment are undergoing or soon will be undergoing clinical evaluation and selection of appropriate patients for these trials is of great importance.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of cervix cancer
2. A decision to treat using radiation therapy according to the existing treatment policies of the PMH Gynecology Group
3. Clinical stage IB-IV with grossly evident cervical disease
4. No distant metastases
5. No cytotoxic anti-cancer therapy for cervical carcinoma prior to study entry
6. Signed informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2006-08-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
To understand the mechanisms by which hypoxia and IFP influence disease progression, and response to radiotherapy, chemotherapy and other novel biologically-targeted therapies in patients with cervix cancer. | 3 months during the first two years, every 4-6 months during years 3 to 5 and yearly thereafter.

SECONDARY OUTCOMES:
To determine if tissue biomarkers of hypoxia are independent prognostic factors for relapse and survival in patients with cervix cancer. | 3 months during the first two years, every 4-6 months during years 3 to 5 and yearly thereafter.
To determine if plasma biomarkers of hypoxia are independent prognostic factors for relapse and survival in patients with cervix cancer. | 3 months during the first two years, every 4-6 months during years 3 to 5 and yearly thereafter.
To assess the heterogeneity of tissue biomarkers of hypoxia in multiple biopsies from cervix cancers. | 3 months during the first two years, every 4-6 months during years 3 to 5 and yearly thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fyles, MD, Principal Investigator — University Health Network, Princess Margaret Hospital; Michael Milosevic, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada